CLINICAL TRIAL: NCT01416805
Title: Utilizing Health Information Technology to Improve Health Care Quality: Implementation of a Computerized Cognitive Behavioral Therapy Protocol for Childhood Anxiety
Brief Title: Computerized Cognitive Behavioral Therapy for Childhood Anxiety in Community Health Centers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Access Behavioral Health (Other); Henderson Behavioral Health (Unknown); Directions for Mental Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R18HS018665 (AHRQ)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-03

CONDITIONS: Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder
Keywords: childhood anxiety disorders; cognitive behavioral therapy; CBT; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder; Psychotherapy; Counseling; Social Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Computerized Cognitive Behavioral Therapy
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavioral Therapy — Those who choose to participate will be enrolled in the 14 week study (18 weeks for phase II). They will required to attend 3 assessments - pre-treatment (week 0), mid-treatment (week 8), and post-treatment (week 14) (and a 4th assessment for a 1 month Follow-up for Phase II at week 18). This group will follow the CCBT protocol (Camp Cope-A-lot), which is the computer-assisted intervention for anxious children being examined in this study. The first 6 levels of this program are skill building levels to be completed by the user in his/her own home. The remaining 6 levels are completed with the therapist and consist of exposure tasks and rehearsal geared toward each child.
  Arms: Computerized Cognitive Behavioral Therapy
Behavioral: Treatment as usual — Those who choose to participate will be enrolled in the 14 week study (18 weeks for phase II). They will required to attend 3 assessments - pre-treatment (week 0), mid-treatment (week 8), and post-treatment (week 14) (and a 4th assessment for a 1 month Follow-up for Phase II at week 18). Those in this group will not receive the CCBT, and instead will undergo therapy for their anxiety as they usually would, whether by using medication or working with a therapist.
  Arms: Treatment as Usual

SUMMARY:
This study will examine the efficacy of a computerized cognitive behavioral therapy (CCBT) program for children with anxiety disorders in community health centers. The first phase of the study will offer insight into the feasibility of providing this intervention in community health centers, while the second phase will compare CCBT to treatment as usual.

DETAILED DESCRIPTION:
Childhood anxiety disorders are quite common and associated with significant psychosocial impairment and distress. Offering equivalent efficacy to pharmacotherapy without the common side effect profile, cognitive behavioral therapy (CBT) is a first line treatment for anxiety disorders in youth. However, dissemination of CBT to community settings is very limited. Effective treatment via traditional CBT often necessitates that the patient travel to a center that specializes in this treatment, and cost can prove an impediment to those of lower socioeconomic status, in particular. As well, differing theoretical approaches and training result in a minority of children with anxiety receiving evidence-based CBT. Accordingly, there is a great need for more widely accessible practices. As such, we are proposing a two phase trial that evaluates the feasibility of implementing a patient-centered intervention in community mental health centers, followed by an efficacy trial. In Phase I, an open trial of computerized CBT (CCBT) will be completed that focuses on feasibility issues of providing this intervention in community mental health centers. Thereafter, we will complete a randomized controlled trial comparing CCBT to treatment as usual (TAU) in Phase II. The open trial will recruit 18 youth ages 7 to 13 years, with the purpose of testing both practicality and management of an already developed CCBT protocol (Kendall & Khanna, 2008). The outcome trial will recruit 110 youth, with the purpose of measuring the efficacy of the CCBT protocol in front-line settings. Significantly greater symptom reductions in the CCBT group as compared to the TAU group would provide critical evidence for the inclusion of CCBT as a treatment option for anxious youth without immediate access to such in-person care. While this study will be coordinated by the University of South Florida Rothman Center for Neuropsychiatry team who is located at All Children's Hospital (USF/ACH), recruitment will take place at three community mental health centers throughout Florida that serve families of lower socioeconomic status. Primary outcomes will be assessed by an independent evaluator, and will include change in anxiety symptom severity; response rates; and remission rates. CCBT will follow the Kendall and Khanna (2008) manual with appropriate integrity checks. The implications of this study are significant, as computerized CBT may enable widespread dissemination of efficacious therapy for anxiety disorders among youth.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient boys and girls with an anxiety disorder (see below) aged 7-13 years.
* Meets DSM-IV criteria for a diagnosis of one of the following anxiety disorders: separation anxiety disorder (SAD), generalized anxiety disorder (GAD), or social phobia.
* Minimum score of 14 on the PARS Severity Scale.
* The child has a Full Scale IQ greater than 80 as assessed on the Wechsler Abbreviated Scale of Intelligence.
* Have home access to a computer with internet connection.

Exclusion Criteria:

* Receiving concurrent psychotherapy or other counseling services.
* New Treatments: Initiation of an antidepressant within 12 weeks before study enrollment or an antipsychotic 6 weeks before study enrollment. No new alternative medications, nutritionals or therapeutic diets within 6 weeks of study enrollment. However, pharmacological interventions may be initiated or added if the child is randomized to the Treatment as Usual arm in Phase II.
* Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxiolytics) within 8 weeks before study enrollment (6 weeks for antipsychotic). Alternative medications that might have behavioral effects must be stable for 6 weeks prior to the study baseline assessment. Any medications that the child is on must remain stable during treatment unless s/he is randomized to the Treatment as Usual arm in Phase II.
* (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months.
* Lifetime DSM-IV bipolar disorder, schizophrenia, or schizoaffective disorder.
* Unwillingness of parents to make the commitment to accompany their children for study visits/assessments.
* Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Storch, Ph.D., Principal Investigator — University of South Florida
Locations (4):
- United States (4):
  - Directions for Mental Health, Clearwater, Florida
  - Henderson Behavioral Health, Fort Lauderdale, Florida
  - Access Behavioral Health, Pensacola, Florida
  - Eric Storch, Tampa, Florida

REFERENCES:
- [Derived] Smarason O, Guzick AG, Goodman WK, Salloum A, Storch EA. Predictors and Moderators of Treatment Outcomes for Anxious Children Randomized to Computer-Assisted Cognitive Behavioral Therapy or Standard Community Care. J Child Adolesc Psychopharmacol. 2023 Oct;33(8):316-324. doi: 10.1089/cap.2023.0019. PMID 37861988
- [Derived] Storch EA, Salloum A, King MA, Crawford EA, Andel R, McBride NM, Lewin AB. A RANDOMIZED CONTROLLED TRIAL IN COMMUNITY MENTAL HEALTH CENTERS OF COMPUTER-ASSISTED COGNITIVE BEHAVIORAL THERAPY VERSUS TREATMENT AS USUAL FOR CHILDREN WITH ANXIETY. Depress Anxiety. 2015 Nov;32(11):843-52. doi: 10.1002/da.22399. Epub 2015 Sep 14. PMID 26366886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computerized Cognitive Behavioral Therapy | Treatment as Usual
Started | 49 | 51
Completed | 45 | 47
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computerized Cognitive Behavioral Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 51 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.8) | 10.2 (1.8) | 9.82 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 26 | 30 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 43 | 41 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: PARS
Description: Pediatric Anxiety Rating Scale (PARS)- The PARS (RUPP, 2002) is a clinician-rated scale assessing anxiety symptoms and the associated severity and impairment in children over the past week. The scale score ranges from 0 to 30 with higher scores reflecting worse anxiety. The score, ranging from 0-30 represents a total score by summing all 6 items (which have item response options ranking from 0 to 5 each).
Time Frame: 14 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computerized Cognitive Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 49 | 51
units on a scale | 11.4 (5.2) | 14.7 (4.9)

2. Secondary Outcome: ADIS-C/P Clinical Severity Rating
Description: Anxiety Disorders Interview Schedule for DSM-IV: Child and Parent Versions (ADIS-IV-C/P)- The ADIS-IV-C/P (Silverman & Albano, 1996) is a clinician-administered, semi-structured interview that assesses for the presence and severity of DSM-IV anxiety disorders as well as Dysthymia and Major Depression, ADHD, Conduct Disorder, and Oppositional-Defiant Disorder. Excellent psychometric properties have been reported (e.g., Wood et al., 2002). The Clinical Severity Rating score is a one item metric reflecting the severity of the anxiety diagnosis. This is rated by the clinician based on their interview with the patient and parent, together with their judgment. The Rating ranges from 0 to 8 with higher scores reflecting worse anxiety.
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computerized Cognitive Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 49 | 51
units on a scale | 3 (1.3) | 4 (1.4)

ADVERSE EVENTS:
Arm/Group | Computerized Cognitive Behavioral Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

LIMITATIONS AND CAVEATS:
The majority of the sample was Caucasian. Not everyone in Treatment as Usual received active treatment. The 1-month follow-up duration was not sufficient to evaluate long-term treatment maintenance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No